CLINICAL TRIAL: NCT01950312
Title: An Open-label Study of the Effects of Gevokizumab in Corticosteroid-resistant Subjects With Autoimmune Inner Ear Disease
Brief Title: The Effects of Gevokizumab in Corticosteroid-resistant Subjects With Autoimmune Inner Ear Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: XOMA (US) LLC (Industry)
Collaborators: Feinstein Institute for Medical Research (Other); National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: X052180; R33DC011827 (NIH)
Record Dates: First submitted 2013-09-20; First posted 2013-09-25 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-02

CONDITIONS: Autoimmune Inner Ear Disease
Keywords: Autoimmune Inner Ear Disease; Inner Ear Disease; Meniere's Disease; Sudden Sensorineural Hearing Loss
MeSH Terms: conditions — Labyrinth Diseases; Meniere Disease; Hearing Loss, Sudden | interventions — gevokizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- gevokizumab (Experimental): Solution for subcutaneous injection
  Interventions: Drug: gevokizumab

INTERVENTIONS:
Drug: gevokizumab

SUMMARY:
The purpose of this study is to determine if gevokizumab therapy may be an alternate therapy in patients with steroid resistant Autoimmune Inner Ear Disease.

ELIGIBILITY:
Inclusion Criteria:

* Autoimmune Inner Ear Disease with active deterioration in at least one ear
* Failure to respond to a trial of high-dose corticosteroid therapy
* Contraceptive measures adequate to prevent pregnancy during the study

Exclusion Criteria:

* Evidence of retrocochlear pathology (vestibular schwannoma) or inner ear malformation (Mondini Malformation or Enlarged Vestibular Aqueduct)
* History of active or chronic infections
* Currently receiving, or having received treatment for a malignancy in the past three years
* Hearing loss that coincides with significant, disabling episodes of vertigo
* History of allergic or anaphylactic reactions to monoclonal antibodies
* Female subjects who are pregnant, planning to become pregnant, have recently delivered, or are breast-feeding

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2013-08; Primary Completion 2015-10 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Improved hearing threshold, as defined by an improvement in either the PTA (Pure Tone Average) of >=5 dB (Decibel), or 12% in the WRS (Word Recognition Score) | Day 28 to Day 84

CONTACTS AND LOCATIONS:
Locations (1):
- Long Island Jewish Medical Center, Hearing & Speech Center, New Hyde Park, New York, United States